CLINICAL TRIAL: NCT03241862
Title: Assess the Impact of Lip Rejuvenation With Restylane® Silk on Projected First Impressions and Mood Perceptions
Brief Title: Assess the Impact of Lip Rejuvenation on Projected First Impressions and Mood Perceptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DeNova Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Silk-FI-01
Record Dates: First submitted 2015-09-14; First posted 2017-08-08 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Lip Rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restylane® Silk (Experimental): All subjects enrolled in the study will undergo lip rejuvenation treatment with Restylane® Silk.
  Interventions: Device: Restylane® Silk

INTERVENTIONS:
Device: Restylane® Silk — Restylane® Silk (Galderma Laboratories, L.P.) is a hyaluronic acid injectable filler, which is approved by the FDA for submucosal implantation for lip augmentation and dermal implantation for correction of perioral rhytids.

SUMMARY:
20 subjects with mild to severe oral commissures or none to severe perioral lines will be enrolled and injected with Restylane® Silk. Photographs will be taken prior to and 14 days after Optimal Cosmetic Results has been achieved, as judged by the investigator.

Changes in the projected first impression will be assessed by a total of 200 blinded evaluators rating the photographs of subjects from the baseline and from 14 days post achieving the Optimal Cosmetic Results. Changes in subjects' mood will be self-assessed through Subjective Happiness Scale and Happiness Measures questionnaires. Aesthetic alterations will be assessed by the investigator via the Global Aesthetic Improvement Scale, Oral Commissure Severity Scale, and the Perioral Lines Severity Scale as well as by the self-assessment of subjects using the Global Aesthetic Improvement Scale.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult of at least 21 years of age;
* Subject has mild to severe oral commissures or none to severe perioral lines, as assessed by the treating investigator;
* Subject is willing and able to provide written informed consent prior to the performance of any study related procedure;
* Subject is willing and able to comply with the protocol requirements; and
* Subject is willing and able to provide written photo consent and adhere to the photography and video procedures such as removal of jewelry and makeup

Exclusion Criteria:

* Subjects who have received lip filler treatments in the past 12 months or neurotoxin injections in the past 6 months;
* Subjects who plan to undergo neurotoxin treatments, ablative skin treatments, facial cosmetic surgery, or other injectable filler treatments during the course of the study;
* Subjects with a known allergy or sensitivity to any component of the study ingredients;
* Subjects with a history of bleeding disorders;
* Female subjects who are pregnant or nursing as well as those who are of childbearing potential but do not employ adequate birth control methods;
* Subjects with severe allergies manifested by a history of anaphylaxis or presence of multiple severe allergies;
* Subjects with previous history of sensitivity to amide type local anesthetics;
* Current history of chronic drug or alcohol abuse;
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study product;
* Subjects who, in the investigator's opinion, have a history of poor cooperation, non-compliance with medical treatment, or unreliability; and
* Enrollment in any active study involving the use of investigational devices or drugs.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Dayan, MD, Principal Investigator — DeNova Research
Locations (1):
- DeNova Research, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restylane® Silk
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Restylane® Silk
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: First Impressions
Description: The projected first impressions are assessed by blinded evaluators using photographs.
  The projected first impressions are assessed by blinded evaluators using the First Impression Questionnaire (FIQ).
  Each of the below First Impression Questionnaire (FIQ) categories is scored between 1 (disagree)-10 (agree) and a total of 8 categories (see below) are assessed for a total possible score of 80. All scores will be graded out of a total possible score of 80 points Social skills Academic Performance Dating Success Occupational success Attractiveness Financial Success Relationship success Athletic success Total scores closer to 80 indicate a more favorable outcome.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: lips first impressions
Arm/Group | Restylane® Silk
Number analyzed (Participants) | 20
Number analyzed (lips first impressions) | 20
score on a scale
  Social skills | 46.756 (0.052)
  Academic Performance | 27.769 (0.887)
  Dating success | 46.391 (0.648)
  Occupational success | 34.404 (0.555)
  Attractiveness | 49.612 (0.544)
  Financial success | 25.029 (0.758)
  Relationship success | 34.245 (0.931)
  Athletic success | 45.433 (0.835)

2. Secondary Outcome: Appearance of the Lip and Perioral Area
Description: Changes in the appearance of the lip and the perioral area are assessed by the PI using the Oral Commissure Severity Scale (OCSS) at Visit 1 and Visit 3/4
  Oral Commissure Severity Scale (OCSS): graded from None (0), Mild (1), Moderate (2), Severe (3)
  None: No wrinkle or fold; slight upturned commissures Mild: Shallow, just perceptible wrinkle or crease; horizontal or slightly downturned corners Moderate: Moderately deep and/or long wrinkle or crease; downturned corners Severe: Very deep and/or long wrinkle or crease; frown at rest
Time Frame: Visit 1 at Baseline and Visit 3 (Week 4) or Visit 4 (Week 6)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restylane® Silk
Number analyzed (Participants) | 20
units on a scale
  Visit 1 | 2.39 (0.502)
  Visit 3/4 | 0.71 (0.470)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Restylane® Silk
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03241862/Prot_SAP_000.pdf